CLINICAL TRIAL: NCT00224835
Title: Mindfulness-Based Stress Reduction and Myocardial Ischemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 319; R01HL072059 (NIH)
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Arteriosclerosis
MeSH Terms: conditions — Arteriosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Mindfulness Based Stress Reduction Class
  Interventions: Behavioral: Mindfulness Based Stress Reduction Class
- 2 (Experimental): Cardiac Education Class
  Interventions: Behavioral: Cardiac Education Class

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction Class — Subjects randomized to this condition will attend 120 minute weekly sessions, plus a 7 hour retreat, for training in mindfulness meditation methods.
  Arms: 1
Behavioral: Cardiac Education Class — Subjects in the disease education control condition will attend 8 weekly 60 minute sessions, plus a 7 hour "special experience" session, all of which will provide information about CAD in a didactic format.
  Arms: 2

SUMMARY:
The principal objective of the study is to evaluate the effectiveness of a widely used complementary medicine intervention, mindfulness-based stress reduction (MBSR), in which mindfulness meditation and yoga are the principal components in the treatment of a chronic, often fatal illness that affects tens of millions of Americans. The investigators propose to conduct a single center randomized controlled trial in which 150 patients will be assigned to either a mindfulness meditation condition, a disease education control condition, or a stress-monitoring usual care control condition. They will test the following specific hypotheses:

1. In comparison to either of the control conditions, significantly more coronary artery disease (CAD) patients in the mindfulness meditation condition will demonstrate reductions in mental stress-induced ischemia.
2. The ratio of low-to-high frequency of spectral power in heart rate variability during ambulatory monitoring will be significantly decreased following the participation in a stress reduction program compared with those in a disease education or usual care condition.
3. Patients in the mindfulness meditation condition will report greater improvement in quality of life (i.e., reductions in general psychological symptomology, anger, anxiety, depression, and daily stress, along with increases in optimism and stress coping efficacy) than patients in either of the control conditions.
4. Day-to-day variability in self-reported mental stress will be inversely related to day-to-day stress coping efficacy in the entire sample and time spent in mindfulness practice in the active treatment condition, and these relationships will be maintained over a 3-month follow-up.
5. Patients with CAD and mental stress ischemia who show an *abnormal peripheral artery response during baseline studies will show a significant improvement after mindfulness intervention.

   * Abnormal responses will be defined as peripheral arterial tonometry (PAT) tracings that decrease greater than 20% in amplitude during mental stress.

DETAILED DESCRIPTION:
BACKGROUND:

Acute and chronic psychological stress has been shown to be a risk factor for cardiac events. More recently with the advent of new technology allowing cardiac imaging, acute psychological stressors have been shown to produce myocardial ischemia in certain subsets of patients with CAD. Several studies have shown that the production of myocardial ischemia in response to acute psychological stress in the laboratory is a marker for adverse events in patients with CAD. Several pathways by which psychologically induced stress may trigger ischemic events have been proposed, and a number of studies have provided evidence that stress affects ischemic events via these pathways. Stress interventions have been shown to have a positive impact on CAD outcomes, with only one thus far testing their effects on ischemic events. Furthermore, some studies have reported positive results with coronary risk factors using meditation and yoga. Current clinical meditation literature suggests that a mindfulness meditation-based stress reduction program (i.e., multicomponent, psychoeducational program based in mindfulness meditation that cultivates an ability to pay attention to one's moment-to-moment experiences in a nonjudgmental, nonreactive fashion) will be able to reduce stress reactivity in CAD patients. It is predicted that such reductions in stress reactivity will result in reduced radionuclide imaged perfusion defects during a laboratory mental stress task. Although it has not been used with heart patients, it has demonstrated good results with both stress and symptomology in the general and other medical populations. We believe that similar results will be seen in CAD patients with effects acting through the following pathways: 1) decreased sympathetic tone and 2) increased parasympathetic tone. The overall goal of the proposed study is to evaluate the efficacy of a meditation-based stress reduction program for the reduction of mental stress-induced ischemia.

DESIGN NARRATIVE:

To test the efficacy of MBSR, patients will be randomly assigned to one of three groups. The MBSR condition will be provided training in mindfulness meditation methods. The patient education control group will be provided information about CAD in a didactic format. This condition will control for the nonspecific effects of contact in a therapeutic setting. Excluding intervals spent in personal meditation practice in the mindfulness meditation condition, the length of sessions in the two intervention conditions will be approximately equal. The third group, a stress-monitoring usual care control condition, will control for the effects of symptom measurement reactivity in patients receiving routine medical care.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Confirmed CAD--the clinical diagnosis of coronary disease will be defined by the presence of at least one of the following: 1) abnormal coronary angiogram; 2) abnormal intravascular ultrasound (IVUS); or 3) abnormal flow reserve and documentation of one of the following: 1) elevated troponin laboratory values typical for myocardial infarction; 2) electrocardiogram (ECG) that shows q-wave abnormalities; 3) nuclear scan that demonstrates a fixed wall motion abnormality consistent with an old myocardial infarct; 4) greater than 95% probability of coronary disease according to the criteria of Diamond and Forrester.102; 5) radionuclide study, dobutamine, or exercise echocardiographic study consistent with stress-induced ischemia (development of segmental wall motion abnormalities or reversible perfusion defects on radionuclide imaging and/or wall motion or systolic thickening abnormalities on stress echocardiographic exam)

Exclusion Criteria:

* Current pregnancy or probability of pregnancy during the duration of the 12-week study
* Diagnosis of unstable angina in the prior 2 months
* Presence of other severe, complicating medical problems that will significantly shorten the patients' life expectancy such that they will not be expected to live for the 12 weeks of this study
* Presence of serious psychopathology evidenced by BDI scores that indicate a clinically critical level of depression (score of 24 or above) with suicidal ideation; previous diagnosis of an organic mental disorder, schizophrenia, or any psychotic disorder; or psychiatric inpatient at any time during the last 5 years (if patients are excluded on the basis of depression scores indicating severe depression or suicidal ideation, referral for psychological services will be offered)
* Post-traumatic stress disorder (PTSD) greater than the 30% VA disability assignment (patients with less severe PTSD will be encouraged to participate)
* Existing meditation practice
* Weight more than 400 pounds

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Psychological stress-induced ischemia (measured by radionuclide imaging at Week 9) | After data collection is complete.
Heart rate variability (measured by AECG at Week 9) | After data collection is complete
Peripheral artery response (measured by finger plethysmography at Week 9) | After data collection is complete
Psychological functioning (degree of depression measured by Beck Depression Inventory (BDI), anxiety by STAI, hostility by Cook-Medley Index, anger by STAXI, optimism by LOT-R, and quality of life/functional status by SF-36 at Weeks 9 and 20) | Results of BDI will be assessed immediately after the participant completes the form. All other questionnaires will be assessed after data collection is complete.
Daily mood diaries (obtained at Weeks 7-8 and Weeks 20-21) | After data collection is complete

CONTACTS AND LOCATIONS:
Overall Officials: David S Sheps, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States